CLINICAL TRIAL: NCT03807349
Title: N-Force Screws Augmented With N-Force Blue in Intracapsular Proximal Femur Fracture Treatment
Brief Title: N-Force Screws Augmented With N-Force Blue in Hip Fractures
Acronym: N-Force
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor will not pursue CE mark for this product, which precludes need for large PMCF study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2017-60T
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Intracapsular Proximal Femur Fracture; Garden Grade I Subcapital Fracture of Femoral Neck; Garden Grade II Subcapital Fracture of Femoral Neck
Keywords: Cannulated Screws; Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- N-Force Screws (Other): N-Force Screws augmented with N-Force Blue in Intracapsular Femur Fractures.
  Interventions: Device: N-Force Screws Augmented with N-Force Blue

INTERVENTIONS:
Device: N-Force Screws Augmented with N-Force Blue — N-Force Fixation System 7.3 mm (Non-fenestrated/fenestrated) applied with washers; N-Force Blue (Bone Substitute Material)

SUMMARY:
The objective of this prospective study is to confirm safety and performance of N-Force Screws augmented with N-Force Blue applied in intracapsular proximal femur fracture treatment.

DETAILED DESCRIPTION:
Primary Endpoint:

• Re-operation within 12 months after initial surgery to promote fracture healing, relieve pain, treat infection, or improve function.

Secondary Endpoints:

* Radiographic and clinical fracture healing of the proximal femur using standard scoring methods and patient satisfaction.
* Cost effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patient has primary Garden I or II intracapsular proximal femur fracture requiring surgical intervention and is eligible for fixation by three cannulated screws augmented with N-Force Blue.
* Patient receives operative treatment within 7 days of injury.
* Patient was ambulatory before injury.
* Patient is 50 years of age or older.

Exclusion Criteria:

* Patient has Garden III or IV intracapsular proximal femur fracture.
* Patient has major cognitive impairment (including dementia).
* Patient is on dialysis.
* Patient is not expected to survive follow-up schedule.
* Patient is expected to have problems maintaining follow-up compliance, i.e. patients with no fixed address, patients not mentally competent to give informed consent, etc. (Investigator's discretion).
* Patient is a prisoner.
* Patient is known to be pregnant and/or breastfeeding.
* Patient is a known alcohol or drug abuser.
* Patient had previous/has active acute or chronic infections, especially at the site of operation.
* Patient has non-viable bone, or has areas where surrounding bone is not viable or capable of supporting and anchoring the implant.
* Patient has traumatic injuries with open wounds or close to the proximal femur fracture, which are likely to become infected.
* Patient is expected to be non-compliant with recommended post-operative weight-bearing instructions.
* Physical conditions, in the opinion of the investigator, that would prohibit adequate implant support or impede healing.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, MBA, Study Director — Zimmer Biomet
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Washington University, St Louis, Missouri
  - Donald B Slocum Research and Education Foundation, Eugene, Oregon
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Force Screws
Started | 12
Completed | 3
Not Completed | 9
Not completed — Early Study Termination | 9

BASELINE CHARACTERISTICS:
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 77 [54 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reoperation
Description: Reoperation after initial surgery to promote fracture healing, relieve pain, treat infection, or improve function.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Number of Participants With Radiographic Fracture Healing of the Intracapsular Femur (RUSH)
Description: Radiographic fracture healing as seen on x-ray and defined using Radiographic Union Score for Hips (RUSH) scoring system. The RUSH quantifies four measures of healing: cortical bridging, cortical fracture disappearance, trabecular consolidation, and trabecular fracture disappearance. Cortical healing is assessed in four anatomic femoral neck regions (anterior, posterior, medial, lateral) and trabecular healing is measured with two assessments (fracture line disappearance and consolidation of matrix). Each of the 10 assessed dimensions of radiographic femoral neck healing are scored 1 to 3, leading to a minimum score of 10 (no signs of healing) and a maximum score of 30 (perfect healing).
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: At the time of early study termination, 12 subjects enrolled into the study. At 6 weeks, data was available for all 12 subjects; at 3 months, data was available for 9 subjects; at 6 months, data was available for 5 subjects; and, at 12 months, data was available for 3 of the 12 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
Participants
  6 weeks - RUSH Healing | 5
  3 months - RUSH Healing: number analyzed (Participants) | 9
  3 months - RUSH Healing | 6
  6 months - RUSH Healing: number analyzed (Participants) | 5
  6 months - RUSH Healing | 5
  12 months - RUSH Healing: number analyzed (Participants) | 3
  12 months - RUSH Healing | 3

3. Secondary Outcome: Participant Steinberg Classification at 12 Months
Description: Steinberg Classification is based on the radiographic appearance and location of lesion. It is concise and delineates the progression and extent of Avascular Necrosis (AVN) involvement more accurately.
  [stage 0:] normal or non-diagnostic radiographs, MRI and bone scan of at risk hip (often contralateral hip involved, or patient has risk factors and hip pain) [stage I:] normal radiograph, abnormal bone scan and/or MRI [stage II:] cystic and sclerotic radiographic changes [stage III:] subchondral lucency or crescent sign [stage IV:] flattening of femoral head, with depression graded into mild: <2 mm moderate: 2-4 mm severe: >4 mm [stage V:] joint space narrowing with or without acetabular involvement [stage VI]: advanced degenerative changes
Time Frame: 12 months
Population: At the time of early study termination, 12 subjects enrolled into the study. Steinberg classification is only measured for subjects that have completed their 12 month follow-up visit. Although 3 subjects completed the 12 month follow-up, Steinberg Classification is only available on 2 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Force Screws
Number analyzed (Participants) | 2
Participants
  Stage 0: Normal radiographs | 1
  Stage VI: Advanced degenerative changes | 1

4. Secondary Outcome: Average FIX-IT Score (Clinical Fracture Healing of the Intracapsular Femur)
Description: The Function IndeX for Trauma (FIX-IT) score is an assessment tool for patients with lower extremity fractures, incorporating pain and the ability to weight-bear. The score utilizes two questions to assess the ability to bear weight and two questions to assess pain at the fracture site. The maximum subtotal for each set of questions is 6 points, yielding a maximum overall score of 12 points and a minimum score (lowest weight bearing and highest pain) of 0 points.
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
score on a scale
  6 week - Fix-IT Score | 6.4 (2.4)
  3 month - Fix-IT Score: number analyzed (Participants) | 9
  3 month - Fix-IT Score | 8.2 (2.1)
  6 month - Fix-IT Score: number analyzed (Participants) | 5
  6 month - Fix-IT Score | 8.6 (3.5)
  12 month - Fix-IT Score: number analyzed (Participants) | 3
  12 month - Fix-IT Score | 7 (5.3)

5. Secondary Outcome: Average EQ-5D-5L Score (Clinical Fracture Healing of the Intracapsular Femur)
Description: The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death.
  The Health Status is scored on a VAS scale of 0 to 100, where 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
score on a scale
  6 week - EQ-5D Score | .605 (.257)
  3 month - EQ-5D Score: number analyzed (Participants) | 9
  3 month - EQ-5D Score | .674 (.136)
  6 month - EQ-5D Score: number analyzed (Participants) | 5
  6 month - EQ-5D Score | .719 (.131)
  12 month - EQ-5D Score: number analyzed (Participants) | 3
  12 month - EQ-5D Score | .542 (.420)
  6 week - Health Status | 68.7 (17.1)
  3 month - Health Status: number analyzed (Participants) | 9
  3 month - Health Status | 74.4 (25.2)
  6 month - Health Status: number analyzed (Participants) | 5
  6 month - Health Status | 68 (23.1)
  12 month - Health Status: number analyzed (Participants) | 3
  12 month - Health Status | 78.3 (2.9)

6. Secondary Outcome: Average Harris Hips Score (Clinical Fracture Healing of the Intracapsular Femur)
Description: This will be measured using Harris Hip Score. This is quantified on a scale of 0-100 and the domains covered are pain, function, absence of deformity, and range of motion. The score is quantified on a scale of 0-100, with 100 points being the best possible outcome. The domains cover pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
score on a scale
  6 weeks - Harris Hip Score | 55.7 (16)
  3 months - Harris Hip Score: number analyzed (Participants) | 9
  3 months - Harris Hip Score | 59.3 (17.6)
  6 months - Harris Hip Score: number analyzed (Participants) | 5
  6 months - Harris Hip Score | 65.4 (15.7)
  12 months - Harris Hip Score: number analyzed (Participants) | 3
  12 months - Harris Hip Score | 68.7 (28.7)

7. Secondary Outcome: Number of Participants That Performed Timed Up-and-Go Test (Clinical Fracture Healing of the Intracapsular Femur)
Description: This will be measured using the Timed 'Up-and-Go' Test. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.This test is used to assess a person's mobility and requires both static and dynamic balance. Scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
Participants
  6 Week - Did Patient perform test? | 5
  3 Month - Did Patient perform test?: number analyzed (Participants) | 9
  3 Month - Did Patient perform test? | 6
  6 Month - Did Patient perform test?: number analyzed (Participants) | 5
  6 Month - Did Patient perform test? | 4
  1 Year - Did Patient perform test?: number analyzed (Participants) | 3
  1 Year - Did Patient perform test? | 1

8. Secondary Outcome: Average Participant Time to Complete Timed Up-and-Go Test (Clinical Fracture Healing of the Intracapsular Femur)
Description: as for outcome 7
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: At the time of early study termination, 12 subjects enrolled into the study. At 6 weeks, data was available for all 12 subjects (only 5 could complete the test); at 3 months, data was available for 9 subjects (only 6 could complete the test); at 6 months, data was available for 5 subjects (only 4 could complete the test); and, at 12 months, data was available for 3 (only 1 could complete the test) of the 12 subjects.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | N-Force Screws
Number analyzed (Participants) | 12
seconds
  6 Week - Average Time to Complete Test (seconds): number analyzed (Participants) | 5
  6 Week - Average Time to Complete Test (seconds) | 21.8 (9.5)
  3 Month - Average Time to Complete Test (seconds): number analyzed (Participants) | 6
  3 Month - Average Time to Complete Test (seconds) | 35.3 (39.9)
  6 Month - Average Time to Complete Test (seconds): number analyzed (Participants) | 4
  6 Month - Average Time to Complete Test (seconds) | 15.5 (7)
  1 Year - Average Time to Complete Test (seconds): number analyzed (Participants) | 1
  1 Year - Average Time to Complete Test (seconds) | 11 (0)

9. Secondary Outcome: Cost-Effective Analysis
Description: Analysis will be performed comparing N-Force to standard non-augmented cannulated screws.
Time Frame: 12 months
Population: Cost effective analysis was not performed due to lack of overall study data.
Arm/Group | N-Force Screws
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Per the protocol, ISO definitions were followed for adverse event data collection. All adverse events were captured for subjects enrolled through 12 months follow-up or study completion (including lost to follow-up), whichever came first.
Description: ISO definition is not materially different from clinicaltrials.gov definitions.
Arm/Group | N-Force Screws
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Force Screws (N=12)
Leg Pain and failure to thrive (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Force Screws (N=12)
Bout of dizziness (Cardiac disorders) | 1
Right knee pain (Musculoskeletal and connective tissue disorders) | 1
Diagnosed with Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Swollen left knee (Musculoskeletal and connective tissue disorders) | 1
Left groin pain (Musculoskeletal and connective tissue disorders) | 1
Lower Extremity/Foot Swollen (Musculoskeletal and connective tissue disorders) | 1
Left hip pain and weakness after multiple falls (Musculoskeletal and connective tissue disorders) | 1
Strike Alert (Nervous system disorders) | 1
Scratched eye from contacts (Eye disorders) | 1
AVN (Musculoskeletal and connective tissue disorders) | 1
Screw loosening (Product Issues) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03807349/Prot_SAP_000.pdf